CLINICAL TRIAL: NCT07220954
Title: A Phase I, Single-Dose, Open-Label, Sequential, Randomised, Crossover Study to Assess the Relative Bioavailability of Different Subcutaneous Formulations of AZD6234 in Participants Living With Overweight or Obesity
Brief Title: A Study to Assess the Relative Bioavailability of Different Subcutaneous Formulations ofAZD6234
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D8750C00008
Record Dates: First submitted 2025-10-23; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: Relative Bioavailability; Pharmacokinetics; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 3 treatment sequences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence ABCD (Experimental): Participants will receive a single SC injection of AZD6234 in each of four study periods, Treatment A in Period 1, Treatment B in Period 2, Treatment C in Period 3 and Treatment D in Period 4 (Where A is AZD6234 Formulation 1, B is AZD6234 Formulation 2 (low concentration), C is AZD6234 Formulation 2 (high concentration) and D is AZD6234 Formulation 3)
  Interventions: Drug: AZD6234 Formulation 1; Drug: AZD6234 Formulation 2 (low concentration); Drug: AZD6234 Formulation 2 (high concentration); Drug: AZD6234 Formulation 3
- Sequence BCAD (Experimental): Participants will receive a single SC injection of AZD6234 in each of four study periods, Treatment B in Period 1, Treatment C in Period 2, Treatment A in Period 3 and Treatment D in Period 4 (Where A is AZD6234 Formulation 1, B is AZD6234 Formulation 2 (low concentration), C is AZD6234 Formulation 2 (high concentration) and D is AZD6234 Formulation 3)
  Interventions: Drug: AZD6234 Formulation 1; Drug: AZD6234 Formulation 2 (low concentration); Drug: AZD6234 Formulation 2 (high concentration); Drug: AZD6234 Formulation 3
- Sequence CABD (Experimental): Participants will receive a single SC injection of AZD6234 in each of four study periods, Treatment C in Period 1, Treatment A in Period 2, Treatment B in Period 3 and Treatment D in Period 4 (Where A is AZD6234 Formulation 1, B is AZD6234 Formulation 2 (low concentration), C is AZD6234 Formulation 2 (high concentration) and D is AZD6234 Formulation 3)
  Interventions: Drug: AZD6234 Formulation 1; Drug: AZD6234 Formulation 2 (low concentration); Drug: AZD6234 Formulation 2 (high concentration); Drug: AZD6234 Formulation 3

INTERVENTIONS:
Drug: AZD6234 Formulation 1 — AZD6234 Formulation 1 will be administered as a single SC injection
  Other Names: AZD6234
Drug: AZD6234 Formulation 2 (low concentration) — AZD6234 Formulation 2 (low concentration) will be administered as a single SC injection
  Other Names: AZD6234
Drug: AZD6234 Formulation 2 (high concentration) — AZD6234 Formulation 2 (high concentration) will be administered as a single SC injection
  Other Names: AZD6234
Drug: AZD6234 Formulation 3 — AZD6234 Formulation 3 will be administered as a single SC injection
  Other Names: AZD6234

SUMMARY:
This study in healthy volunteers aims to compare blood levels and side effects after administration of different formulations of AZD6234.

This study will take place at one site in Nottingham, United Kingdom, and will enrol 21 healthy men and women aged 18-55 years.

DETAILED DESCRIPTION:
This study in healthy volunteers aims to compare blood levels and side effects after administration of different formulations of AZD6234.

This study will take place at one site in Nottingham, United Kingdom.

It plans to enrol 21 healthy men and women aged 18-55 years.

Each volunteer will take part in 4 treatment periods and receive different formulations of AZD6234, by injection under the skin into the abdomen (stomach). In each period they'll be given a single dose without food. They'll stay in the clinic for 6 nights on 4 occasions, attend up to 10 outpatient visits, and take up to 19 weeks to finish the study.

Blood and urine samples will be collected to: measure the amount of AZD6234 and its breakdown products, do safety tests and assess the effect of the test medicine on the immune system response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating females aged 18 to 55 years inclusive
* BMI of 25.0 to 35.0 kg/m2 inclusive and weight ≥50 kg

Exclusion Criteria:

* History of any clinically important disease or disorder
* History or presence of clinically significant cardiovascular, renal, hepatic, dermatological, respiratory, neurological, psychiatric or gastrointestinal disorder including a history of pancreatitis or gall stones
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the planned first dosing day
* Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis
* Any clinically significant abnormal findings in vital signs
* Any clinically significant abnormalities on 12-lead ECG
* HbA1c ≥6.5% (≥48 mmol/mol)
* Evidence of renal impairment
* Females who are pregnant or lactating.
* Any participant who has received an amylin analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer)
* Participants who report to have previously received AZD6234.
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Plasma sample collection from pre- dose to 30 days post final dose
  Assess relative bioavailability (rBA) by comparing the pharmacokinetics (PK) of different AZD6234 SC formulations
Area under the concentration-time curve from time 0 to the time of the last measurable concentration (AUC0-t) | Plasma sample collection from pre- dose to 30 days post final dose
  Assess relative bioavailability (rBA) by comparing the pharmacokinetics (PK) of different AZD6234 SC formulations
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) | Plasma sample collection from pre- dose to 30 days post final dose
  Assess relative bioavailability (rBA) by comparing the pharmacokinetics (PK) of different AZD6234 SC formulations

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs)/serious AEs (SAEs), and change from baseline for vital signs, electrocardiograms (ECGs), and laboratory safety tests | Through study duration, approximately 19 weeks
  Safety and tolerability of different AZD6234 SC formulations
Time of maximum observed plasma concentration (tmax) | Plasma sample collection from pre- dose to 30 days post final dose
  Pharmacokinetics (PK) of different AZD6234 SC formulations
Terminal elimination half-life (t1/2) | Plasma sample collection from pre- dose to 30 days post final dose
  Pharmacokinetics (PK) of different AZD6234 SC formulations
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) | Plasma sample collection from pre- dose to 30 days post final dose
  Pharmacokinetics (PK) of different AZD6234 SC formulations
Volume of distribution based on the terminal phase calculated using AUC0-inf after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) | Plasma sample collection from pre- dose to 30 days post final dose
  Pharmacokinetics (PK) of different AZD6234 SC formulations

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/